CLINICAL TRIAL: NCT06910475
Title: Exerkidney: A Tracking of Uremic Toxins, Exerkines, Genetic Aspects, Physical Fitness, Body Composition, and The Effects of Physical Training in People With Chronic Kidney Disease at Different Stages
Brief Title: Physical Exercise and Biomolecular Analysis to Reduce Uremic Toxins in Chronic Kidney Disease: An Exploratory Study
Acronym: DRC_LExS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of Brasília (Other)
Responsible Party: Principal Investigator, Lysleine Alves de Deus, Principal Investigator, Catholic University of Brasília
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 79266224.1.0000.002979266224.1; 445068/2023-0 (Other Grant/Funding Number: CNPq)
Record Dates: First submitted 2024-10-03; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Kidney Disease, Chronic; Kidney Failure Chronic
Keywords: Exerkines; uremic toxins; physical training; physical exercise; indoxyl sulfate; p-Cresyl sulfate; hippuric acid; trimethylamine N-oxide; asymmetric dimethylarginine; redox balance; inflammation; tumor necrosis factor alpha; interleukin; leptin; irisin; BNDF; ancestry; telomere
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Inflammation | interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Intervention Model Description: The intervention of the study will consist of physical exercise, including aerobic exercise, resistance training, and concurrent training (a combination of both). These interventions will follow a structured and supervised training protocol to assess their effects on the selected outcomes.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Conservative CKD (Experimental): Patients with CKD under conservative treatment.
  Interventions: Other: Resistance training; Other: Endurance training; Other: Concurrent training
- Hemodialysis (Experimental): Patients with CKD under hemodialysis treatment.
  Interventions: Other: Resistance training; Other: Endurance training; Other: Concurrent training
- Peritonial dialysis (Experimental): Patients with CKD under peritonial dialysis.
  Interventions: Other: Resistance training; Other: Endurance training; Other: Concurrent training
- Transplant patient (Experimental): Transplant patient
  Interventions: Other: Resistance training; Other: Endurance training; Other: Concurrent training
- Control group - conservative (No Intervention): Patients with CKD under conservative treatment.
- Control group - Hemodialysis (No Intervention): Pacients under hemodialysis treatment
- Control group - peritonial dialysis (No Intervention): Patients under peritonial dialysis
- Control group - Transplant patient (No Intervention): Transplant patient

INTERVENTIONS:
Other: Resistance training — The training program will follow a periodized approach, starting with a low total volume (loads x sets x repetitions), ensuring gradual adaptation, patient safety, and performance progression. Strength training will begin 48 hours after muscle strength tests.Sessions will occur 2 to 4 times per week on non-consecutive days. Each session will include 6-12 exercises, with 1-3 seconds for concentric and eccentric actions, 6-20 repetitions, 1-6 sets, and 1-3 minutes of rest. Intensity will be gauged by perceived exertion, ranging from "easy" to "hard," with load adjustments every 2 months based on progress.Patients undergoing hemodialysis may perform the sessions during or between treatments. Portable equipment like free weights, ankle weights, and resistance bands will be used.
  Arms: Conservative CKD; Hemodialysis; Peritonial dialysis; Transplant patient
Other: Endurance training — Training sessions will be conducted 2 to 4 times per week on non-consecutive days. Patients will perform aerobic training on different ergometers, namely: bicycle, treadmill, and stair climber. The choice will depend on the patient's needs/abilities and/or equipment availability. The load will be adjusted between 50% and 100% of the ventilatory threshold, according to the patient's cardiorespiratory capacity. The duration of the training will vary between 10 and 60 minutes, always starting with low load and volume, with gradual progression to ensure patient comfort and safety.
  Arms: Conservative CKD; Hemodialysis; Peritonial dialysis; Transplant patient
Other: Concurrent training — Training sessions will be conducted 2 to 6 times per week, alternating between strength training one day and aerobic training the next, as described above. As patients improve their physical fitness, strength and aerobic training may be performed on the same day.
  Arms: Conservative CKD; Hemodialysis; Peritonial dialysis; Transplant patient

SUMMARY:
The accumulation of uremic toxins is detrimental to physiological systems and induces premature biological aging. Renal function assessment methods, such as predictive formulas, may be influenced by ancestry in Brazilians, given the country's ethnic diversity, resulting in inaccurate estimates. On the other hand, physical exercise is an important ally in treating chronic kidney disease (CKD) as it induces metabolic changes that help slow the disease's progression. Additionally, the anti-aging effect conferred on those who engage in physical exercise is widely recognized. However, investigations into the impact of physical exercise on the concentration of uremic toxins and biological aging in patients with chronic kidney disease and their relationship with ancestry are still in the early stages and inconclusive. The investigators aim to track uremic toxins, exerkines, genetic aspects, nutritional profile, physical fitness, body composition, and the effects of different types of physical training (periodized and progressive) in people with chronic kidney disease at various stages. Additionally, to verify associations between these factors and their effects on different physiological systems. This is a triple-blind randomized clinical trial, with a 10-year follow-up of patients. The sampling will be non-probabilistic in terms of accessibility or convenience. Adult volunteers of both biological sexes aged 18 or older, with chronic kidney disease in conservative treatment (stages 2, 3, 4, and 5, n~400), patients undergoing renal replacement therapy (hemodialysis or peritoneal dialysis, n~800), and transplant recipients (n~400) will be recruited from different hemodialysis centers. After being grouped by disease stage, patients will be randomized according to pre-training variables and then allocated to the following groups: control group (CTL; at least n~100), strength training (ST; at least n~100), aerobic training (AT; at least n~100), and combined training (CT; at least n~100). The patients will undergo evaluations of body composition, cardiorespiratory capacity, muscle strength, autonomic nervous system function, and nutritional, psychological, and biomolecular assessments. The training protocols will be adjusted according to the patient's physical capacity, always considering periodization and progression.

DETAILED DESCRIPTION:
This study is a randomized, triple-blind clinical trial with a 10-year follow-up. Sampling is non-probabilistic by accessibility or convenience. Recruitment: Recruitment will be widely promoted via mass media (social media, TV) to invite individuals with chronic kidney disease. Additionally, the investigators will receive referrals from partner physicians and public-private partnerships. Participants will be recruited from dialysis clinics, outpatient clinics, and hospitals in Brasília, DF, respecting privacy and confidentiality. The investigators aim to recruit a minimum of 1,600 adult patients (both sexes), aged 18+, divided into those with CKD in conservative treatment (stages 2, 3, 4, 5, n~400), renal replacement therapy (hemodialysis and peritoneal dialysis, n~800), and kidney transplant patients (n~400). Participants will receive all pertinent information about the study and potential risks and benefits. Those who agree will sign an informed consent form. Following consent, each patient will undergo a comprehensive history assessment, including exercise, medical, and nutritional histories, along with an analysis of their medical records. Monthly evaluations will cover all procedures and interventions outlined for their allocated group. Patient Randomization: Participants will be stratified by CKD stage (conservative treatment, hemodialysis, peritoneal dialysis, and post-transplant) and further randomized by pre-training variables (biological sex, body weight, BMI, and body composition), using an online application. Patients will then be allocated to one of four groups: control (CTL; n~100), strength training (ST; n~100), aerobic training (AT; n~100), and combined training (CT; n~100). Assessments: Body Composition: BMI, DEXA, 7-Skinfold (Jackson and Pollock protocol); Cardiopulmonary Capacity: Anaerobic threshold, Fitcheck, respiratory muscle strength, spirometry; Muscle Strength: 1RM, handgrip, isokinetic force and power, E-lastic portable dynamometer; Autonomic Nervous System: Cardiovascular regulation during deep breathing, Valsalva maneuver with handgrip exercise, post-exercise ischemia, cold-water hand immersion, perceived exertion, respiratory rate, heart rate, arterial oxygen saturation, HRV, BPV, spontaneous baroreflex sensitivity, EEG, cognitive assessment; Nutritional Assessment: 24-hour dietary recall, food frequency questionnaire; Psychological Assessment: Quality of life (KDQOL-SF36), sleep quality, Beck Depression Inventory; Biochemical and biomolecular Assessments: Biological sample collection (urine, feces, saliva, blood) for measurements of creatinine, cystatin-C, leptin, GDF-15, TGF-β, insulin, albumin, SIRT-1, C-reactive protein, irisin, intact FGF23, C-terminal FGF23, ADMA, soluble α-Klotho, glycated hemoglobin (HbA1c), total cholesterol, LDL-c, HDL-c, triglycerides, myeloperoxidase, lipoperoxidation assay, paraoxonase-1, total antioxidant capacity, nitric oxide, lactate, creatine kinase, uremic toxins (KIM-1, NGAL, indoxyl sulfate, p-cresyl sulfate, TMAO, TNF-α, IL-6, ADMA, exercise-related proteins, BDNF, DNA and RNA isolation (salting out method), telomere length and telomerase activity, microRNA expression analysis, HPLC quantification, and identification of compounds by MALDI TOF/TOF mass spectrometry); Ancestry Analysis: Ancestry genome-wide association stratification; Training Protocols: Physical training protocols will include strength, aerobic, and combined training; Statistical Analysis: Sample size is calculated for 99% power (1-β = 0.99) with an alpha of 5% (α = 0.05) and effect size of 0.1, resulting in 400 patients. Descriptive analysis will be presented in tables and charts. Normality and homogeneity of data will be tested by Shapiro-Wilk and Levene's tests. For normally distributed data, group comparisons will be conducted by two-way ANOVA with Tukey's post-hoc test for significant differences. Non-normally distributed data will be analyzed by Kruskal-Wallis with Dunn's post-test, with results expressed as medians and interquartile ranges. Significance will be set at p < 0.05, with effect size calculated by Cohen's d. Associations between variables will be evaluated by Spearman's correlation. To minimize type II error, the investigators will calculate variations before and after training as Δ = post-training - pre-training. Principal Component Analysis (PCA) and individual variability analysis will use delta results to identify key variables affecting estimated glomerular filtration rate. This analysis will use the Past software (v4.09). Typical error and smallest worthwhile change (SWC) will be calculated per Swinton et al. (2018). Effect size will follow Hopkins' scale: <0.2 (trivial), 0.2-0.6 (small), 0.6-1.2 (moderate), 1.2-2.0 (large), 2.0-4.0 (very large), >4.0 (extremely large). Additionally, K-means cluster analysis, an unsupervised machine learning method, will identify patterns based on numerical distance between variables. Statistical analyses will use Microsoft Excel® 2010, GraphPad Prism 6.0, R and RStudio (v4.1.3), and SPSS (v.21.0).

ELIGIBILITY:
Inclusion Criteria:

* those diagnosed with chronic kidney disease and presenting persistent albuminuria (>300mg/g) following KDIGO guidelines;
* metabolic syndrome {i.e., type 2 diabetes mellitus, arterial hypertension (blood pressure >180/100mmHg), overweight or obesity, and dyslipidemia};
* no complications arising from pre-existing clinical metabolic diseases (i.e., diabetic coma, ketoacidosis, hyperosmolarity, and/or uncontrolled diabetes), as evaluated by a nephrologist;
* absence of neurodegenerative, musculoskeletal, lupus erythematosus, or congenital kidney disease;
* no apparent cardiovascular complications, such as heart failure, severe arrhythmia, angina, or cerebrovascular disease;
* no comorbidities that limit performance in physical tests or training;
* not engaged in exercise programs for at least six months prior to the start of the experimental protocol;
* no smoking or alcohol consumption behavior;
* D-dimer values within normal range (220-500 ng/mL FEU)

Exclusion Criteria:

* regularly engage in physical exercise,
* have suffered a stroke in the last 6 months and/or present autoimmune diseases,
* have unstable cardiac dysfunctions, such as: uncontrolled coronary artery disease, aneurysm at risk of rupture, uncontrolled arrhythmia, uncontrolled hypertension (SBP > 190 mmHg and/or DBP > 100 mmHg), heart attack in the last 3 months;
* infectious conditions, Hb < 8 in the last routine monthly hemodialysis exam;
* musculoskeletal pain;
* fever;
* resting SpO2 lower than 94%;
* restriction by the clinical team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female
Enrollment: 1600 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentrations of uremic toxins - Indoxyl sulfate | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum concentration of Indoxyl sulfate (µmol/L) will be measured.
Concentrations of uremic toxins - p-Cresyl sulfate | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum concentration of p-Cresyl sulfate (µmol/L) will be measured.
Concentrations of uremic toxins - hippuric acid | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum concentration of hippuric acid (µmol/L) will be measured.
Concentrations of uremic toxins - trimethylamine N-oxide | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum concentration of trimethylamine N-oxide (µmol/L) will be measured.
Concentrations of uremic toxins - screening | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Other uremic toxins may also be identified through miRNA expression, high-performance liquid chromatography (HPLC) and mass spectrometry (MALDI TOF/TOF) identified peptides, with spectra processed via FlexControl and FlexAnalysis.
Serum albumin | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  The serum albumin (mg/dL) will be measured in duplicate using the automated chemical analyzer (COBAS c111 system, Roche Diagnostics, Switzerland).
Creatinine | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Creatinine (mg/dL) will be measured in duplicate using the automated chemical analyzer (COBAS c111 system, Roche Diagnostics, Switzerland).
Cystatin C levels | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Cystatin C levels (mg/dL) will be measured in duplicate using the automated chemical analyzer (COBAS c111 system, Roche Diagnostics, Switzerland).
Estimation of renal function in patients undergoing conservative treatment | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  The values of creatinine and cystatin C values will be applied to the formula proposed by Inker (2012) to estimate the glomerular filtration rate (eGFR).

SECONDARY OUTCOMES:
Anthropometric measures - weight | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Weight in kilograms.
Cardiopulmonary capacity - Graded Incremental Test and Metalyzer 3B | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Graded Incremental Test: Conducted on a cycle ergometer with a stepped or ramped protocol, ECG is monitored for abnormalities by a cardiologist. Gas exchange (VE, VO₂, VCO₂ L/min) is measured using the Metalyzer 3B gas analyzer (Cortex Biophysik) calibrated with a 3L syringe, and mixed gas (4.9% CO₂, 17% O₂). Values are recorded during the last 20 seconds of each 3-minute stage. The anaerobic threshold is determined by VE/VO₂ (L/min) and VE/VCO₂ (L/min) ratios.
Autonomic function - Cardiovascular Autonomic Regulation during Deep Breathing | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Patients should breathe deeply and slowly in sync with the rhythm of a metronome, completing one respiratory cycle every 10 seconds (i.e., respiratory rate = 6 cycles/min). The maneuver will be conducted for 1 minute and 20 seconds, corresponding to 8 respiratory cycles. After a 5-minute rest interval, the maneuver will be repeated. The highest heart rate during each inspiration will be subtracted from the lowest heart rate during the subsequent expiration. The average of the five largest responses will be used to interpret the heart rate response to deep breathing, which serves as a marker of cardiac vagal control.
Nutritional profile - dietary recall | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Nutritional assessment will use a 24-hour dietary recall to determine each patient's average intake of food and nutrients. Detailed data on types and amounts (in grams) of foods consumed will be collected, allowing calculations of proteins, lipids, cholesterol, carbohydrates, fiber, vitamins, and minerals. Dietary Reference Intakes will be used to evaluate dietary adequacy, and data will be analyzed with the Webdiet Health Manager application.
Telomere length | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Average telomere length will be measured in monocytes. Telomere length will be assessed using quantitative real-time PCR (qPCR) using specific primers. Electrophoresis and Quantification: Amplification products will be analyzed using agarose gel electrophoresis with ethidium bromide. Bands (~300 base pairs) will be quantified by densitometry using Image J® software, with standardized background enhancement and a fixed quadrant dimension.
Exerkinas - serum levels of irisin | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of irisin (ng/mL) will be measured pré and post-training using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Glycemic profile - fasting glucose | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of fasting glucose (mg/dL) will be mesure using the automated chemical analyzer (COBAS c111 system, Roche Diagnostics, Switzerland).
Patient's quality of life | Every two months, over a follow-up period of at least 6 months and up to up to 10 years.
  Kidney Disease and Quality-of-Life Short Form (KDQOL-SF36): This questionnaire has 36 items across eight general health dimensions: physical functioning, limitations from physical health, emotional health, social functioning, mental health, pain, vitality, general health perception, and current health status vs. one year ago. The kidney-specific section includes eleven dimensions: symptoms/problems, effects on daily life, burden, work status, cognitive function, social interactions, sexual function, sleep, social support, dialysis staff encouragement, and patient satisfaction . The scoring procedure first transforms the raw precoded numeric values of items to the 0-100 possible range, with higher transformed scores always reflecting a better quality of life. Then, the items scale is averaged together to create the scale scores. The results of each scale vary from 0 to 100 (worst to best possible status).
Gut microbiota profile | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Patients will perform self-collection following the instructions provided in the OMNIgene•GUT kit (OMR-200). Instructions will be available through an educational video and a step-by-step guide. Samples will be homogenized and aliquots will be stored in Eppendorf tubes. Samples will be analyzed within three months of collection, following the manufacturer's instructions (DNA Genotek, Ottawa, Ontario, Canada).
Inflammatory profile - TNF-α, IL-6, IL-10, IL-11, IL-18 e FGF-23 | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Inflammatory profile: tumor necrosis factor-alpha (TNF-α), interleukin-6 (IL-6) , interleukin-10 (IL-10), interleukin-11 (IL-11), interleukin-18 (IL-18), Fibroblast Growth Factor 23 (FGF-23) all in pg/mL will be measured using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Ancestry Assessment | Every two months, over a follow-up period of at least 6 months and up to 10 ye Every two months, over a follow-up period of at least 6 months and up to 10 years.ars.
  Genomic analysis will use DNA extracted from participants' blood samples. Genome-wide association studies (GWAS) will be applied to gather ancestry-related data, enhancing the precision of assessing ancestry's influence on renal function. Genome-Wide Association Ancestry Stratification: Ancestry analysis will be based on genetic and phenotypic data, performed by an external company to ensure result quality and reliability. GWAS techniques will identify genetic markers linked to various ancestral origins using blood-derived DNA. CD Genomics, a company specializing in genomic sequencing and genetic data analysis, will conduct the GWAS. The goal is to identify genetic variants associated with renal function across different stages of chronic kidney disease (CKD), incorporating participants' ancestry factors.
Muscle strength - 1-repetition maximum | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Muscle strength will be evaluated through 1-repetition maximum (1-RM), expressed in kilograms-force (kgf)."
Anthropometric measures - height | Every two months, over a follow-up period of at least 6 months and up to up to 10 years.
  Height in meters
Anthropometric measures - Body mass index | Every two months, over a follow-up period of at least 6 months and up to up to 10 years.
  Weight (kg) and height (m) will be combined to report BMI in kg/m².
Body composition - DEXA | Every two months, over a follow-up period of at least 6 months and up to up to 10 years.
  Body composition will also be measured via Dual-energy X-ray Absorptiometry (DEXA) using a GE Lunar Prodigy® (GE Healthcare, Madison, WI, USA) with software version 4.7e. Measurements will be taken with patients fasting for 8+ hours.
Body composition - 7 Skinfold | Every two months, over a follow-up period of at least 6 months and up to up to 10 years.
  The Jackson and Pollock 7-Skinfold Protocol will also be used to estimate body density ( in millimeters) on skinfold measurements at seven body sites: biceps, triceps, subscapularis, suprailiac, middle axillary, abdomen, thigh, and leg. The value of measures will be applied to the equation proposed by Jackson and Pollock and converted to fat percentage based on the equation by Siri (1961).
Psychosocial aspects of patients | Every two months, over a follow-up period of at least 6 months and up to up to 10 years.
  Beck Depression Inventory: This tool has 21 groups of self-evaluative statements (0-3) regarding symptom severity. Scores of 0-9 = no depression, 10-15 = mild, 16-23 = moderate, and 24+ = severe depression.
Cardiopulmonary capacity - Fitcheck | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Fitcheck: The classic graded IT consists of 3-4 stages of 3 minutes each, with 1-minute pauses and 10-watt increases. Gas exchange (VE, VO₂, VCO₂ L/min) is assessed via Fitcheck® (Brazil, 2022), and this test is performed intra- and inter-dialysis for renal patients. The anaerobic threshold is determined by VE/VO₂ (L/min) and VE/VCO₂ (L/min) ratios.
Cardiopulmonary capacity - Respiratory Muscle Strength | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Respiratory Muscle Strength: Pimax and Pemax are measured with a digital manovacuometer (MVD300-U Homed®) using nasal clips and oral adapters per ATS/ERS (2002). Spirometry: Conducted with Contec SP8B, measures (L/min) FVC, FEV1, FEV1/FVC, FEF25/75, FEF25/75/FVC seated, per ATS/ERS.
Autonomic function - Valsalva Maneuver | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  The Valsalva maneuver will be used to induce sudden and significant changes in blood pressure, enabling the assessment of heart rate, blood pressure, and muscle sympathetic nerve activity responses. The maneuver will be performed in the supine position. Patients will perform an expiratory effort for 15 seconds, maintaining an expiratory pressure of approximately 40 mmHg. The maneuver will be repeated two to three times, with at least a 10-minute interval between attempts, to enhance the reliability of the results.
Autonomic function - Handgrip Exercise | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  The maximum voluntary contraction will be determined as the highest force value obtained from three reproducible attempts. During these attempts, participants will be instructed to increase force abruptly and maintain a plateau for 2 to 3 seconds. The maximum force value will be used to calculate 30% of this value, which must be sustained for 2 minutes. During the exercise, the force trace will be projected onto the ceiling to help participants maintain the target force value as established in the protocol.
Autonomic function - Post-Exercise Ischemia | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Circulatory occlusion will be performed by inflating a cuff positioned on the proximal portion of the arm. The occlusion will be applied before the end of the exercise to ensure that the metabolites produced during the exercise remain trapped in the arm, maintaining the activation of metaboreceptors even after exercise cessation.
Autonomic function - Cold pressure test | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Cold exposure will be conducted by immersing one hand in a container filled with ice water. This maneuver activates pain receptors, which in turn provoke an increase in sympathetic activity. Therefore, this test will provide a means to assess the effect of increased sympathetic activity per se on the peripheral chemoreflex, independently of muscle metaboreflex activation.
Autonomic function - handgrip strenght | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Handgrip strength ( kgf) will be measured using a digital force transducer specifically designed for this type of exercise (Grip Force Transducer, ADInstruments).
Autonomic function - respiratory rate | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Respiratory rate will be measured using a belt positioned on the lower portion of the thorax. This belt will monitor the expansion and contraction of the thoracic cavity during the respiratory cycle, allowing for precise measurement of respiratory rate (Piezo Respiratory Belt Transducer, ADInstruments). Respiratory rate, tidal volume, minute volume, end-tidal partial pressure of oxygen (PETO₂), and end-tidal partial pressure of carbon dioxide (PETCO₂) will be measured on a breath-by-breath basis using a metabolic analyzer (CPX Ultima, MedGraphics). The analyzer will be calibrated before each experiment following the manufacturer's instructions.
Autonomic function - Heart rate | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Heart rate will be calculated from the electrocardiogram (ECG) signal, which will be measured using a single lead configuration (3 Lead Bio Amp Cable, ADInstruments). Also, heart rate will be measured using a three-lead electrocardiogram (Finometer, Finapres) for integration of simultaneous recordings to simultaneously record the various assessed variables on the same timescale, a system for converting analog signals to digital signals will be used (Powerlab, ADInstruments).
Autonomic function - Arterial Oxygen Saturation | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Arterial oxygen saturation will be measured using an oximeter positioned on the earlobe (Oximeter Pod/Ear Clip, ADInstruments).
Autonomic function - blood pressure | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Blood Pressure: Beat-to-beat blood pressure will be measured using the photoplethysmography method, with an appropriately sized cuff positioned on the middle finger of the non-dominant hand (Finometer, Finapres).
Autonomic function - Femoral Artery Measurements | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  The diameter of the femoral artery and blood flow velocity will be assessed using Doppler ultrasound (Vivid 7, GE).
Autonomic function - Heart Rate Variability (HRV) | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  HRV will be analyzed in time and frequency domains.
Autonomic function - Spontaneous Baroreflex Sensitivity (SBS) | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  The analysis of spontaneous baroreflex sensitivity will be performed using two methods: cross-spectral analysis and sequence analysis. Cross-spectral analysis will consist of calculating the square root of the ratio between the LF band power of HRV and the LF band power of SAP. Sequence analysis will involve identifying sequences of three or more consecutive beats where an increase/decrease in SAP is followed by an increase/decrease in the RR interval. This variable is largely determined by the vagal branch of the autonomic nervous system.
Autonomic function - Instantaneous Cerebral Electrical Activity | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Instantaneous cerebral electrical activity will be assessed using the NeuroVirtual - Humanizing Diagnostics BWIII EEG Plus with 36 channels, following the 10-20 system and frequency adjustments through the equipment's application. The procedures will be conducted in accordance with the manufacturer's instructions.
Nutritional profile - Food Frequency Questionnaire | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Food intake will also be assessed with the Food Frequency Questionnaire for hemodialysis patients (FFQ-HD), covering eleven food groups, including grains, vegetables, legumes, fruits, meats, dairy, oils, seasonings, beverages, sweets, and canned foods. Frequency and quantity over the past 12 months will be estimated, aided by a photo album for portion reference.
Exerkinas - adiponectin | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of adiponectin (µg/mL) will be measured pre and post-training using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Exerkinas - α-Klotho and sirtuin-1 (SIRT-1) | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of α-Klotho (pg/mL) and sirtunin - SIRT-1 (pg/mL) will be measured pre and post-training using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Exerkinas - Sestrin | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of sestrin (ng/mL) will be measured pré and post-training using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Exerkines - screening | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Additional exercise-related biomarkers will be screened through HPLC and identified by MALDI TOF/TOF MS (Bruker). Peptides and their purity will be assessed, and spectra will be analyzed using FlexControl 3.4 and FlexAnalysis 3.4.
Glicemic profile - glycated hemoglobin | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of glycated hemoglobin (mmol/mol) will be mesure using the automated chemical analyzer (COBAS c111 system, Roche Diagnostics, Switzerland).
Glycemic profile - insulin | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of insulin (pmol/L) will be mesure using the automated chemical analyzer (COBAS c111 system, Roche Diagnostics, Switzerland).
Glycemic profile - HOMA-IR | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  The HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) is used to estimate insulin resistance based on fasting glucose and insulin levels. The values of fasting glucose and fasting insulin are applied in the following formula: Fasting Insulin(μU/mL)×Fasting Glucose(mg/dL)/405.
Glycemic profile - HOMA-B | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  The HOMA-B (Homeostatic Model Assessment for Beta-Cell Function) is used to estimate pancreatic beta-cell function based on fasting glucose and insulin levels. It helps assess how well the pancreas is producing insulin in response to blood glucose levels.The formula for HOMA-B is: Fasting Insulin(μU/mL)×360 /Fasting Insulin(μU/mL)×360.
Lipid profile | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Total cholesterol (mg/dL), cHDL(mg/dL), cLDL (mg/dL), and triglycerides (mg/dL) will be measured using the automated chemical analyzer (COBAS c111 system, Roche Diagnostics, Switzerland).
Inflammatory profile - CRP | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of C-reactive protein (CRP; mg/L) will be mesured using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Inflammatory profile - MPO, Leptin, GDF-15 | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of myeloperoxidase (MPO), leptin, Growth/differentiation factor 15 (GDF-15) all in ng/mL will be mesured using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Inflammatory profile - ADMA | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of Asymmetric Dimethylarginine (ADMA; µmol/L) will be mesured using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Redox profile - TBARS e NOx | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of Thiobarbituric acid reactive substances (TBARS) and nitric oxide (NOx) all in µmol/L will be mesured using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Redox balance - paraoxonase-1 and catalase | Every two months, over a follow-up period of at least 6 months and up to Every two months, over a follow-up period of at least 6 months and up to 10 years.10 years.
  Serum levels of paraoxonase-1 and catalase (all in U/mL) will be mesured using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Redox profile - TROLOX | : Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of total antioxidant capacity (µmol Trolox Eq/L) wil be mesured using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Redox balance - SOD | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Serum levels of superoxide dismutase (SOD; U/mg protein) will be mesured using Human Enzyme-Linked Immunosorbent Assay (ELISA) Kit.
Telomerase Activity Measurement | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Telomerase activity will be measured in monocytes. Telomerase activity will be evaluated via the Telomeric Repeat Amplification Protocol (TRAP). RT-PCR for TRF1, TRF2, and POT1: To identify TRF1, TRF2, and POT1 genes, a Reverse Transcriptase reaction followed by PCR will be conducted using specific primers. Electrophoresis and Quantification: Amplification products will be analyzed using agarose gel electrophoresis with ethidium bromide. Bands (~300 base pairs) will be quantified by densitometry using Image J® software, with standardized background enhancement and a fixed quadrant dimension.
Muscle strength - handgrip | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Muscle strength will be evaluated through handgrip dynamometry, expressed in kilograms-force (kgf).
Muscle strength - isokinetic dynamometry | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Muscle strength will be evaluated through isokinetic dynamometry, expressed in kilograms-force (kgf).
Muscle strength - e-lastic | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Muscle strength will be evaluated through e-lastic, portable dynamometry, expressed in kilograms-force (kgf).
Autonomic function - Stroke Volume | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Stroke volume will be estimated using the Modelflow method.
Autonomic function - Cardiac Output | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  Cardiac Output and Peripheral Vascular Resistance: These will be calculated based on the estimated stroke volume.
Autonomic function - Blood Pressure Variability (BPV) | Every two months, over a follow-up period of at least 6 months and up to 10 years.
  BPV will be analyzed in time and frequency domains.

CONTACTS AND LOCATIONS:
Overall Officials: Thiago S Rosa, PhD, Principal Investigator — Catholic University of Brasília; Hugo L Correa, MSc, Study Chair — Catholic University of Brasília
Locations (1):
- Catholic University of Brasília, Taguatinga, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No